CLINICAL TRIAL: NCT07135102
Title: A Clinical Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of [225Ac]Ac-PSMA-XT Injection in Patients With Metastatic Castration-resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xiaorong Sun (Other)
Responsible Party: Sponsor-Investigator, Xiaorong Sun, Director of Nuclear Medicine Department, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2024-365-01
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 225Ac-PSMA-XT treatment (Experimental)
  Interventions: Drug: 225Ac-PSMA-XT

INTERVENTIONS:
Drug: 225Ac-PSMA-XT — Patients will receive 225Ac-PSMA-XT administration at an interval of 6 weeks between each dose.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of 225Ac -labeled PSMA ligand(PSMA-XT) in the treatment of mCRPC

ELIGIBILITY:
Inclusion Criteria:

1. have the ability to understand and sign an approved informed consent form (ICF).
2. >= 18 years old.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. have a life expectancy >6 months.
5. have histological, pathological, and/or cytological confirmation of prostate cancer.
6. PSMA Positron Emission Tomography (PET)/Computed Tomography (CT) scan positive
7. have a castrate level of serum/plasma testosterone (<50 ng/dL or <1.7 nmol/L).
8. have received at least one NAAD (such as enzalutamide and/or abiraterone)； patients must have been previously treated undergone at least 1-2 prior taxane-based chemotherapy regimens or be unsuitable for taxane therapy (unsuitability includes contraindications, investigator-determined ineligibility, or patient refusal) in mCRPC stage.
9. progressive mCRPC.
10. have adequate organ function。
11. Subjects of childbearing potential voluntarily use an effective method of contraception, such as condoms, oral or injectable contraceptives, Intra-uterine device（IUD）,etc., during treatment and within 6 months of the last use of the trial drug.

Exclusion Criteria:

1. Previous treatment with any of the following within 6 months of enrollment: Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, hemi-body irradiation. Previous PSMA-targeted radioligand therapy is not allowed.

   Known other malignancies.
2. Any systemic anti-cancer therapy (e.g. chemotherapy, immunotherapy or biological therapy within 28 days prior to day of enrollment.
3. Known hypersensitivity to the components of the study therapy or its analogs.
4. A superscan as seen in the baseline bone scan.
5. Patients with a history of Central Nervous System (CNS) metastases.
6. Uncontrolled, intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, cardiac arrhythmia, or other severe complications.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events | Through study completion, assessed up to 2 years
  To evaluate the safety and tolerability of [177Lu]Lu-PSMA-XT Injection assessed from the number and incidence of patients with adverse events using CTCAE v5.0 and physical examination, electrocardiogram and laboratory abnormality, etc.
Dose-limiting toxicity（DLT） | Through study completion, assessed up to 2 years
  Incidence and severity of dose-limiting toxicities.

SECONDARY OUTCOMES:
Prostate-specific Antigen 50 (PSA50) Response | Through study completion, assessed up to 2 years.
  PSA50 response was defined as the proportion of participants who had a >= 50% decrease in PSA from baseline confirmed by a PSA measurement >= 4 weeks later.
Radiographic Progression-free Survival (rPFS) | Through study completion, assessed up to 2 years.
  Radiographic progression-free survival (rPFS) was defined as the time (in months) from the date of enrollment to the date of radiographic disease progression per the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria or death due to any cause.
Overall Response Rate (ORR) | Through study completion, assessed up to 2 years.
  Overall Response Rate (ORR) was defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR). ORR was based on RECIST 1.1 response for patients with measurable disease at baseline.
Duration of Response (DOR) | Through study completion, assessed up to 2 years.
  Duration of Response (DOR) was defined as the duration between the date of first documented Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) and the date of first documented radiographic progression or death due to any cause .
Disease Control Rate (DCR) | Through study completion, assessed up to 2 years.
  Disease control rate (DCR) was defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) according to RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Shandong First Medical University, Jinan, Shandong, China